CLINICAL TRIAL: NCT03364127
Title: Double-blind Phase 2 RCT: Effect of Acupuncture on Patient Vulvodynia Outcomes
Brief Title: Effect of Acupuncture on Patient Vulvodynia Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Judith Schlaeger, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-0885
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Vulvodynia; Vulvodynia, Generalized; Vulvar Vestibulitis
Keywords: Vulvar Pain, Dyspareunia
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis; Dyspareunia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Active Acupuncture (Active Comparator): Active Acupuncture two times per week for 5 weeks
  Interventions: Other: Active Acupuncture
- Placebo Acupuncture (Placebo Comparator): Placebo Acupuncture two times per week for 5 weeks
  Interventions: Other: Placebo Acupuncture

INTERVENTIONS:
Other: Active Acupuncture — Active Acupuncture two times per week for 5 weeks
  Other Names: Penetrating Acupuncture Needle
  Arms: Experimental: Active Acupuncture
Other: Placebo Acupuncture — Placebo Acupuncture two times per week for 5 weeks
  Other Names: Skin-touch Placebo Needle
  Arms: Placebo Acupuncture

SUMMARY:
This study evaluates acupuncture for the treatment of vulvodynia; specifically if it reduces vulvar pain and pain with intercourse. It also examines how long the effect of acupuncture lasts in women with vulvodynia. Half of the women will receive acupuncture and the other half will receive placebo acupuncture. Women who get a reduction in pain will monitor there pain once a week for up to 12 weeks to see how long the acupuncture effect lasts.

DETAILED DESCRIPTION:
The investigators' goal is to demonstrate the effects of acupuncture for the treatment of vulvodynia. Up to 14 million American women have vulvodynia, a debilitating pain syndrome characterized by pain (burning, irritation, stinging or rawness) in the vulva and dyspareunia that renders sexual intercourse virtually impossible and leaves these women desperate for relief. Not only are women in pain, but they often lose their partners or have relationship difficulties due to their inability to have sexual intercourse. No therapies have been proven efficacious and rapid pain relief is unpredictable and rarely possible. After exhausting Western Medicine options, these women often turn to acupuncture. But in contrast to other pain conditions, there have been no acupuncture sham control studies of vulvodynia.

Only four studies, including one of the investigators', provide some evidence of the effect of acupuncture on vulvodynia. In three, single-group acupuncture studies, women had less pain, better quality of life, improved sexual health, and improved mental health. The investigators' randomized wait-list controlled pilot study of 36 women with vulvodynia showed great promise. The investigators found a statistically significant and clinically meaningful reduction in vulvar pain and dyspareunia, and an increase in overall sexual function after a 5-week, 13-needle, 10 session acupuncture protocol. This newly developed, standardized acupuncture treatment protocol is the first breakthrough in the treatment of this puzzling disorder. It includes acupuncture points that relieve pain in the genitals. The results of the investigators' initial pilot study provided the first evidence from a two-group design that the acupuncture protocol could reduce pain intensity, pain during intercourse, and increase overall sexual function. These findings, however, warrant stronger evidence to support the inference that the effect is indeed due to the acupuncture since ours or no other study included a sham control or provided follow-up data beyond immediate posttest, which means that the duration of the acupuncture effect is unknown. The investigators' recent feasibility study paves the way to overcome this gap by use of double-blind acupuncture needles. Findings from these two studies support the investigators' proposal for the world's first double-blind randomized controlled trial (RCT) of acupuncture for vulvodynia while exploring its duration of effect.

The investigators propose a phase 2 double-blind, pretest/posttest RCT to compare effects of penetrating needles or the skin touch placebo needles on vulvar pain in our 13-needle, 10-session acupuncture treatment protocol. A sample of 130 women, with a diagnosis of vulvodynia, either generalized or provoked vestibulodynia, 18 to 45 years of age will be recruited from clinical and community settings and 80 subjects are expected to complete the study. Stratified by type of vulvodynia, participants will be randomized 1:1 either to the penetrating needle group or the skin touch placebo needle group. These double-blind needles will provide a strong sham procedure to mask both the acupuncturist and subject to the type of needle used for the 10-treatment protocol.

Specific aims are to:

Aim 1. Compare the penetrating needle group and the skin touch placebo needle group for effects on the: (a) primary outcome: vulvar pain (PAINReportIt® average pain intensity, 0-10), and (b) secondary outcomes: dyspareunia (FSFI dyspareunia) and sexual function (FSFI total). The investigators hypothesize that controlling for baseline values, at posttest there will be statistically significant less vulvar pain (primary) and dyspareunia and better sexual function in the penetrating needle group compared to the skin touch placebo group.

Aim 2. In participants with a clinically meaningful reduction in pain intensity (at least 1.5 points) at posttest compared to pretest, describe the duration of the acupuncture treatment and placebo effects weekly until pain returns to pretest or up to 12 weeks after posttest. The investigators will describe the variability over time in vulvar pain intensity (0-10) after a tampon insertion-removal stimulus and thereby explore the duration of the effect by intervention group, vulvodynia subgroups, and demographic subgroups (e.g., age, race, occupation). These findings will provide insights to guide future research on initial and maintenance acupuncture for vulvodynia.

ELIGIBILITY:
Inclusion Criteria:

1. a previous diagnosis of generalized vulvodynia or provoked vestibulodynia
2. 18 to 45 years old
3. a pain now score 4 or higher with tampon insertion and removal performed at the initial screening exam
4. speak and read English

Exclusionary Criteria:

1. infectious conditions of the vulva/vagina
2. inflammatory conditions of the vulva/vagina
3. neoplastic disorders of the vulva/vagina
4. neurologic disorders of the vulva/vagina
5. trauma to the genitals
6. iatrogenic conditions of the genitals
7. hormonal deficiencies
8. co-morbid pelvic pain conditions (to avoid confounding pain outcomes) such as pelvic inflammatory disease and documented history of endometriosis
9. menopause

Patients may have a history of but not have active in the last 6 months migraine headaches, temporomandibular joint disease (TMJ), irritable bowel syndrome (IBS), interstitial cystitis, painful bladder syndrome, or fibromyalgia.

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith M. Schlaeger, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago College of Nursing, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The data generated by our research are available from the PI, Judith M. Schlaeger, upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available immediately upon release of this ClinicalTrials.gov website for 5 years.
Access Criteria: Please email the Principal Investigator: Judith Schlaeger, jschlaeg@uic.edu

REFERENCES:
- [Derived] Schlaeger JM, Suarez ML, Glayzer JE, Kobak WH, Meinel M, Steffen AD, Burke LA, Pauls HA, Yao Y, Takayama M, Yajima H, Kaptchuk TJ, Takakura N, Foster D, Wilkie DJ. Protocol for double-blind RCT of acupuncture for vulvodynia. Contemp Clin Trials Commun. 2022 Nov 2;30:101029. doi: 10.1016/j.conctc.2022.101029. eCollection 2022 Dec. PMID 36387991
- [Derived] Desloge AA, Patil CL, Glayzer JE, Suarez ML, Kobak WH, Meinel M, Steffen AD, Burke LA, Yao Y, Takayama M, Yajima H, Kaptchuk TJ, Takakura N, Foster DC, Wilkie DJ, Schlaeger JM. Women's Experience of Living with Vulvodynia Pain: Why They Participated in a Randomized Controlled Trial of Acupuncture. J Integr Complement Med. 2023 Jan;29(1):50-54. doi: 10.1089/jicm.2022.0647. Epub 2022 Sep 21. PMID 36130137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four-hundred and fifty women were assessed for eligibility of which 290 did not meet eligibility criteria and 71 declined to participate. Eighty-nine participants were enrolled between February 2018 and September 2022. Participants were recruited from community settings as well as from medical clinics throughout the Chicagoland area, from healthcare provider referrals, and from the National Vulvodynia Association website.
Pre-assignment Details: No participants were excluded after randomization and assignment to the groups.
Period: Overall Study
Arm/Group | Experimental: Active Acupuncture | Placebo Acupuncture
Started | 45 | 44
Completed | 39 | 42
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Population: The analysis population is the same as the population in Participant Flow.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Active Acupuncture | Placebo Acupuncture | Total
Number analyzed (Participants) | 45 | 44 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.0 (8.25) | 31.4 (8.35) | 30.2 (8.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 34 | 35 | 69
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 31 | 31 | 62
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 6 | 4 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 44 | 89

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Intensity Will be Measured With the Pain Intensity Numbers Scale (PINS).
Description: The subject calls the pain intensity a number ranging between the minimum value, 0 and 10, the maximum value. Zero represents "no pain" and 10 represents"pain as bad as it could be". Higher scores mean more pain. The PINS will include three items (pain now, least and worst pain in the past 24 hours), which are used to calculate the average of pain intensity. The PINS with the three items and standardized instructions is part of PAINReportIt® which is an electronic version of the 1970 version of the McGill Pain Questionnaire.
Time Frame: baseline and after the 10th acupuncture treatment week 5
Population: Participants receiving active acupuncture and placebo acupuncture
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Active Acupuncture | Placebo Acupuncture
Number analyzed (Participants) | 45 | 44
score on a scale
  Baseline | 3.90 (2.39) | 3.51 (2.31)
  After the 10th acupuncture treatment week 5 | 2.48 (2.11) | 2.22 (2.09)
Statistical Analysis 1: Comparison: Experimental: Active Acupuncture vs Placebo Acupuncture; Test type: Superiority; p = 0.702, ANCOVA; Full information maximum likelihood for missing data and to retain participants for intention to treat model. Adjusted for baseline value; Mean Difference (Net) = -.12, 95% CI 2-sided [-.76 to .51]

2. Secondary Outcome: Dyspareunia Subscale of the Female Sexual Function Index (FSFI)
Description: The Dyspareunia Subscale of the FSFI measures pain with sexual intercourse. The FSFI consists of three items scored using a scale ranging from zero to five. The scores of the three items are then summed and multiplied by a factor of 0.4, resulting in a minimum score of 0 and a maximum score of 6.0, with higher scores indicating less pain with sexual intercourse.
Time Frame: baseline and after the 10th acupuncture treatment week 5
Population: Participants receiving active acupuncture and placebo acupuncture.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Active Acupuncture | Placebo Acupuncture
Number analyzed (Participants) | 45 | 44
score on a scale
  Baseline | 1.22 (0.89) | 1.38 (1.16)
  after the 10th acupuncture treatment week 5 | 1.61 (1.76) | 1.83 (1.82)
Statistical Analysis 1: Comparison: Experimental: Active Acupuncture vs Placebo Acupuncture; Test type: Superiority; p = 0.77, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = .10, 95% CI 2-sided [-.58 to .79]

3. Secondary Outcome: Total Score of the Female Sexual Function Index (FSFI)
Description: The FSFI is a 19-item, multi-dimensional, self-report measure that measures overall sexual function from six domains of sexual response: desire, arousal, lubrication, orgasm, satisfaction, and dyspareunia. The six subscale scores are measured on a scale of 0-5 for each item. Individual item responses from each of the 6 domains are added together to achieve a domain score and are each multipled by a factor (desire, 0.6; arousal, 0.3; lubrication, 0.3; orgasm, 0.4; satisfaction, 0.4; and dyspareunia, 0.4). These final domain scores are summed to obtain the Total Score of the FSFI, ranging from 2.0 to 36.0, with higher scores indicating better overall sexual function.
Time Frame: baseline and after the 10th acupuncture treatment week 5
Population: Participants receiving active acupuncture and placebo acupuncture.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental: Active Acupuncture | Placebo Acupuncture
Number analyzed (Participants) | 45 | 44
score on a scale
  Baseline | 15.9 (7.05) | 17.4 (5.92)
  After the 10th acupuncture treatment week 5 | 17.0 (8.29) | 19.3 (7.71)
Statistical Analysis 1: Comparison: Experimental: Active Acupuncture vs Placebo Acupuncture; Test type: Superiority; p = 0.436, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.16, 95% CI 2-sided [-1.76 to 4.09]

4. Secondary Outcome: Vulvar Pain Intensity Will be Measured With the Pain Intensity Numbers Scale (PINS).
Description: The subject calls the pain intensity a number between 0, the minimum value and 10, the maximum value. Zero is "no pain" and 10 is "pain as bad as it could be." Higher scores indicate a worse outcome. The PINS will include one item (vulvar pain intensity). The PINS with vulvar pain intensity and standardized instructions is part of PAINReportIt® which is an electronic version of the 1970 version of the McGill Pain Questionnaire.
Time Frame: after the 10th acupuncture treatment weekly up to 12 weeks post last acupuncture treatment.
Population: Participants receiving active acupuncture and placebo acupuncture that entered the Duration of Effect phase. Participants with a clinically meaningful reduction in pain intensity (at least 1.5 points) at the 10th acupuncture treatment compared to pretest, will measure Vulvar Pain Intensity weekly until pain returns to pretest or up to 12 weeks after the 10th acupuncture treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Experimental: Active Acupuncture/Duration of Effect: Active Acupuncture Duration of Effect measured weekly with Vulvar Pain Intensity post 10th acupuncture treatment weekly up to 12 weeks.
- Placebo Acupuncture/Duration of Effect: Placebo Acupuncture Duration of Effect measured weekly with Vulvar Pain Intensity post 10th acupuncture treatment weekly up to 12 weeks
Arm/Group | Experimental: Active Acupuncture/Duration of Effect | Placebo Acupuncture/Duration of Effect
Number analyzed (Participants) | 24 | 24
score on a scale
  Week 1: number analyzed (Participants) | 18 | 20
  Week 1 | 4.19 (2.33) | 2.60 (2.09)
  Week 2: number analyzed (Participants) | 19 | 22
  Week 2 | 3.37 (2.50) | 3.68 (2.31)
  Week 3: number analyzed (Participants) | 15 | 22
  Week 3 | 3.79 (2.68) | 3.16 (1.98)
  Week 4: number analyzed (Participants) | 13 | 22
  Week 4 | 3.23 (2.09) | 3.23 (2.39)
  Week 5: number analyzed (Participants) | 11 | 16
  Week 5 | 4.55 (2.54) | 3.13 (1.63)
  Week 6: number analyzed (Participants) | 12 | 18
  Week 6 | 3.88 (2.68) | 3.33 (1.78)
  Week 7: number analyzed (Participants) | 9 | 19
  Week 7 | 3.22 (1.99) | 3.84 (2.48)
  Week 8: number analyzed (Participants) | 9 | 17
  Week 8 | 2.67 (1.80) | 2.79 (1.57)
  Week 9: number analyzed (Participants) | 5 | 14
  Week 9 | 4.00 (2.83) | 2.32 (0.99)
  Week 10: number analyzed (Participants) | 10 | 13
  Week 10 | 3.50 (1.78) | 2.77 (1.59)
  Week 11: number analyzed (Participants) | 9 | 14
  Week 11 | 2.89 (2.57) | 3.04 (1.39)
  Week 12: number analyzed (Participants) | 5 | 14
  Week 12 | 5.40 (2.19) | 2.64 (1.22)
Statistical Analysis 1: Comparison: Experimental: Active Acupuncture/Duration of Effect vs Placebo Acupuncture/Duration of Effect; Goal was to assess duration of effect among those who showed a response to the intervention (1.5 or greater decrease in PIN); Test type: Superiority; p = 0.017, Log Rank — Kaplan-Meier curves by treatment arm were examined to determine the rates of return to baseline over the 12-week follow-up period; Hazard Ratio (HR) = 2.72, 95% CI 2-sided [1.13 to 6.54]

ADVERSE EVENTS:
Time Frame: The specific time period over which adverse event data were collected was 5 weeks, which started at the first acupuncture treatment and was completed after the 10th acupuncture treatment.
Description: The definition of adverse events and serious adverse events does not differ from the clinicaltrials.gov definition.
Arm/Group | Experimental: Active Acupuncture | Placebo Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/44
Other Adverse Events (participants affected / at risk) | 0/45 | 0/44

LIMITATIONS AND CAVEATS:
No limitations or caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT03364127/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT03364127/ICF_001.pdf